CLINICAL TRIAL: NCT04023669
Title: St. Jude ELIOT: Phase 1 Evaluation of LY2606368, a Molecularly-Targeted CHK1/2 Inhibitor Therapy, in Combination With Cyclophosphamide or Gemcitabine for Children and Adolescents With Refractory or Recurrent Group 3/Group 4 or SHH Medulloblastoma Brain Tumors
Brief Title: Evaluation of LY2606368 Therapy in Combination With Cyclophosphamide or Gemcitabine for Children and Adolescents With Refractory or Recurrent Group 3/Group 4 or SHH Medulloblastoma Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJELIOT; NCI-2019-04787 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2019-07-11; First posted 2019-07-17 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Brain Tumor; Brain Tumor, Recurrent; Brain Tumor, Refractory; Brain Tumor, Pediatric; Medulloblastoma; Medulloblastoma Recurrent; Medulloblastoma, Non-WNT/Non-SHH; Medulloblastoma, Non-WNT/Non-SHH, Group 3; Medulloblastoma, Non-WNT/Non-SHH, Group 4; Brain Cancer; CNS Cancer; CNS Tumor; CNS Neoplasm
Keywords: Brain Tumors in Adolescents; Brain Tumors in Children; Brain Tumors in Young Adults; CHK1/2 Inhibitor; Combination therapy; Indeterminate molecular subgroup; Medulloblastoma, Group 3; Medulloblastoma, Group 4; Medulloblastoma, G3/G4; Progressive brain tumor; Recurrent brain tumor; Refractory brain tumor; Sonic hedgehog; SHH Medulloblastoma; St. Jude Brain Tumor Studies; St. Jude Studies; St. Jude Treatment; Molecular; Molecular therapy
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma; Central Nervous System Neoplasms; Microphthalmia, Isolated, with Coloboma 5 | interventions — prexasertib; Cyclophosphamide; Gemcitabine; Filgrastim; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A: prexasertib + cyclophosphamide (Experimental): Stratum A: Participants receive combination treatment with cyclophosphamide given intravenously (IV) on days 1 and 15 and prexasertib given intravenously (IV) on days 2 and 16. Cycles repeat every 28 days for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity. They may also receive growth therapy support with filgrastim or peg-filgrastim.
  Note: Only if absolutely necessary, cyclophosphamide may be given on day 16 and prexasertib may be given on day 17.
  Interventions: Drug: Prexasertib; Drug: Cyclophosphamide; Biological: filgrastim; Biological: peg-filgrastim
- B: prexasertib + gemcitabine (Experimental): Stratum B: Participants receive combination treatment with gemcitabine given intravenously (IV) on days 1 and 15 and prexasertib given intravenously (IV) on days 2 and 16. Cycles repeat every 28 days for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity. They may also receive growth therapy support with filgrastim or peg-filgrastim.
  Note: Only if absolutely necessary, gemcitabine may be given on day 16 and prexasertib may be given on day 17.
  Interventions: Drug: Prexasertib; Drug: Gemcitabine; Biological: filgrastim; Biological: peg-filgrastim

INTERVENTIONS:
Drug: Prexasertib — IV
  Other Names: LY2606368
Drug: Cyclophosphamide — IV
  Other Names: Cytoxan
  Arms: A: prexasertib + cyclophosphamide
Drug: Gemcitabine — IV
  Other Names: 2'-deoxy-2',2' difluorocytidine monohydrochloride; LY18801; Gemzar®
  Arms: B: prexasertib + gemcitabine
Biological: filgrastim — Given subcutaneously (SQ). Alternatively, pegfilgrastim may be given.
  Other Names: G-CSF
Biological: peg-filgrastim — Given subcutaneously (SQ). Alternatively, filgrastim may be given.
  Other Names: pegylated filgrastim; PEG filgrastim; Neulasta®

SUMMARY:
SJELIOT is a phase 1 trial that aims to explore the combination of prexasertib with established DNA-damaging agents used in medulloblastoma to evaluate tolerance and pharmacokinetics in recurrent or refractory disease. Additionally, a small expansion cohort will be incorporated into the trial at the combination MTD/RP2D (maximum tolerated dose/recommended phase two dose) to detect a preliminary efficacy signal.

Stratum A: Prexasertib and Cyclophosphamide

Primary Objectives

* To determine the safety and tolerability and estimate the maximum tolerated dose (MTD)/recommended phase 2 dose (RP2D) of combination treatment with prexasertib and cyclophosphamide in participants with recurrent/refractory Group 3 and Group 4 medulloblastoma and recurrent/refractory sonic hedgehog (SHH) medulloblastoma.
* To characterize the pharmacokinetics of prexasertib in combination with cyclophosphamide.

Secondary Objectives

* To estimate the rate and duration of objective response and progression free survival (PFS) associated with prexasertib and cyclophosphamide treatment in this patient population.
* To characterize the pharmacokinetics of cyclophosphamide and metabolites.

Stratum B: Prexasertib and Gemcitabine

Primary Objectives

* To determine the safety and tolerability and estimate the MTD/RP2D of combination treatment with prexasertib and gemcitabine in participants with recurrent/refractory Group 3 and Group 4 medulloblastoma.
* To characterize the pharmacokinetics of prexasertib in combination with gemcitabine.

Secondary Objectives

* To estimate the rate and duration of objective response and PFS associated with prexasertib and gemcitabine treatment in this patient population.
* To characterize the pharmacokinetics of gemcitabine and gemcitabine triphosphate (only at St. Jude Children's Research Hospital).

DETAILED DESCRIPTION:
Participants will be stratified by the biological characteristics of their tumor to one of two treatment strata:

STRATUM A

* Combination Treatment: prexasertib and cyclophosphamide
* Patient population: Participants with recurrent/refractory Group 3 and Group 4 (G3/G4) medulloblastoma, recurrent/refractory sonic hedgehog (SHH) medulloblastoma and medulloblastoma participants with Indeterminate molecular subgroup

STRATUM B

* Combination Treatment: prexasertib and gemcitabine
* Patient population: Participants with recurrent/refractory Group 3 and Group 4 medulloblastoma

Participants with a diagnosis of G3/G4 medulloblastoma who qualify for both treatment strata will be assigned per slot availability as well as institutional PI preference. If slots are available in both stratum A and stratum B, patients will be assigned to the dose level nearest completion.

The Rolling 6 design will be used separately in each stratum to estimate the maximum tolerated dose (MTD) or recommended phase two dose (RP2D). Therapy will be administered in cycles of 28 days and may be continued for up to 24 months (26 cycles) in the absence of disease progression or unacceptable toxicity.

Participants will receive doublet therapy in cycles of 28 days. The dose-limiting toxicity (DLT)-evaluation period will consist of the first cycle until day 1 criteria of cycle 2 has been met. Participants will be evaluated at least once a week during the DLT-evaluation period and at regular intervals thereafter. Standard tests (i.e. physical exams, blood tests, and disease evaluations) will be undertaken at regular intervals. Research-associated evaluations (i.e. pharmacokinetic studies, etc.) will also be carried out during therapy. Treatment may be continued for up to 2 years in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria: Screening Phase

* Participants with recurrent, refractory, or progressive medulloblastoma.
* Age ≥ 1 year and < 25 years at the time of screening.
* Participants and/or guardian can understand and is willing to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria: Screening Phase

* Previous exposure to any CHK1 inhibitor.
* Participants with a history of clinically significant, uncontrolled heart disease and/or repolarization abnormalities.
* Participants with any history of QTc prolongation (i.e. QTc interval of > 480 msec).

Inclusion Criteria: Strata A and B

* Participant must be ≥1 year and <25 years of age at time of screening.
* Participant must have recurrent, progressive or refractory Group 3/Group 4 or SHH medulloblastoma (per central pathology confirmation of primary tissue and/or relapsed tissue). Central pathology review previously completed at St. Jude Children's Research Hospital using equivalent methods can be used for enrollment. Note: Group 3/Group 4 may be referred to as Non-WNT Non-SHH (NWNS) in pathology reports. Medulloblastoma patients with indeterminate molecular subgroup after central pathology review are eligible for enrollment on stratum A.
* Participant must have measurable or evaluable disease as defined in the protocol.
* Participant must have received their last dose of myelosuppressive anticancer chemotherapy at least 3 weeks prior to study enrollment.
* Participants must have had their last fraction of radiation (including CSI) at least 4 weeks prior to study enrollment. Participants who received radiation therapy for palliation must have had their last fraction of radiation at least 2 weeks prior to study enrollment.

  -- Note: Participants must have relapsed with recurrent, progressive or refractory disease after any prior radiation therapy that is not considered palliative. Palliative radiation therapy is defined as local small port RT to alleviate and/or palliate symptoms. (CSI, whole brain RT, large field/port RT, or large field/port multilevel spinal RT will not be considered palliative at any dose.)
* Participant who are receiving corticosteroids must be on a stable or decreasing dose for at least 1 week prior to enrollment with no plans for escalation.
* Participant must have a Lansky (≤ 16 years) or Karnofsky (> 16 years) performance score of ≥50 and, in the opinion of the investigator, a minimum life expectancy of at least 6 weeks.

  -- Note: Participants who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Participant must have adequate bone marrow and organ function as defined as:

  * ANC ≥ 1.0 x 10^9/L without growth factor support within 7 days
  * Platelet count ≥ 75x 10^9/L without support of a platelet transfusion within 7 days
  * Hemoglobin ≥8.0 g/dL without support of a blood transfusion within 7 days
  * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within institutional normal limits or corrected to within normal limits with supplements before first dose of study medication
  * Serum creatinine ≤ the maximum serum creatinine based on age/gender: Age: 1 to < 2 years; maximum serum creatinine (mg/dL): 0.6 (male, female); Age: 2 to < 6 years; maximum serum creatinine (mg/dL): 0.8 (male, female); Age: 6 to < 10 years; maximum serum creatinine (mg/dL): 1 (male, female); Age: 10 to < 13 years; maximum serum creatinine (mg/dL): 1.2 (male, female); Age: 13 to < 16 years; maximum serum creatinine (mg/dL): 1.5 (male), 1.4 (female); Age :≥ 16 years; maximum serum creatinine (mg/dL): 1.7 (male), 1.4 (female).
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 x ULN. For the purposes of this study the ULN of ALT and AST is 45 U/L.
  * Total bilirubin ≤ ULN; or if > ULN then direct bilirubin ≤ 1.5 x ULN
* Female participants of childbearing age must have a negative pregnancy test at the time of enrollment.
* Participants of childbearing or child fathering potential must be willing to use medically acceptable form of birth control during treatment and for 16 weeks after stopping treatment.
* Participants and/or guardian have the ability to understand and the willingness to sign a written informed consent document according to institutional guidelines.

Exclusion Criteria: Strata A and B

* Participant who is receiving any other investigational agents.
* Participants with other clinically significant medical disorders (i.e. serious infections or significant cardiac, pulmonary, hepatic, psychiatric, or other organ dysfunction) that could compromise their ability to tolerate protocol therapy or would interfere with the study procedures or results.
* Participant with a history of clinically significant, uncontrolled heart disease and/or repolarization abnormalities as documented by a standard 12-lead ECG.
* Shortening fraction of <27% by ECHO or ejection fraction of <50% by gated radionuclide study.
* Prior history of QTc prolongation or QTc interval of > 480 msec.
* Female participants who are breastfeeding a child.
* Participants are excluded if unable to comply with guidelines listed in appendix I.

Ages: 1 Year to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-08-08 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2025-01-13 (Actual)

PRIMARY OUTCOMES:
Estimate the Maximum tolerated dose (MTD)/Recommended Phase 2 Dose (RP2D) of each doublet by stratum | 1 month after start of prexasertib and cyclophosphamide or gemcitabine treatment
  The maximum tolerated dose (MTD) is empirically defined as the highest dose level at which six patients have been treated with at most one patient experiencing a dose-limiting toxicity (DLT) and the next higher dose level has been determined to be too toxic. The MTD estimate will not be available if the lowest dose level studied is too toxic or the highest dose level studied is considered safe. In the latter case, the highest studied safe dose may be considered as the recommended phase 2 dose (RP2D). The MTD estimation will be limited to evaluable patients and toxicity assessments from course 1 (28 days).
To determine the safety and tolerability of combination treatment with prexasertib and cyclophosphamide or gemcitabine. | Up to 2 years after start of prexasertib and cyclophosphamide or gemcitabine treatment
  Incidence of adverse event data at least possibly related to treatment will be summarized in tables by treatment combination and by dose level.
To characterize the area under the concentration-time curve (AUC0-∞) of prexasertib in combination with cyclophosphamide or gemcitabine. | prexasertib and cyclophosphamide or gemcitabine treatment course 1 days 2 through 7
  Prexasertib area under the curve (AUC0-∞) is estimated based on course 1, days 2 through 7 PK samples.
To characterize the systemic clearance (CL) of prexasertib in combination with cyclophosphamide or gemcitabine. | prexasertib and cyclophosphamide or gemcitabine treatment course 1 days 2 through 7
  Prexasertib systemic clearance (CL) is estimated based on course 1, days 2 through 7 pharmacokinetic samples.

SECONDARY OUTCOMES:
Rate of objective response (complete or partial response) by stratum | Up to 1 year after completion of prexasertib and cyclophosphamide or gemcitabine treatment
  The incidence of objective responses (complete or partial response) observed during prexasertib and cyclophosphamide or gemcitabine treatment or during follow-up prior to progression or initiation of alternative cancer therapy.
Duration of objective response by stratum | Up to 1 year after completion of prexasertib and cyclophosphamide or gemcitabine treatment
  The duration of objective response is measured from the time the measurement criteria are met for complete response (CR) or partial response (PR), whichever is recorded first, until the first day on which recurrent or progressive disease is objectively documented.
Progression-free survival for patients treated with prexasertib and cyclophosphamide or gemcitabine | Up to 3 years from diagnosis
  Progression-free survival (PFS) is defined from the time of treatment initiation until disease progression or until death from any cause (whichever is earlier) for patients who experience an event and until the date of last follow-up for those who are alive and progression free at the time of analysis. PFS is estimated by Kaplan-Meier approach and median PFS is reported.
To characterize the area under the concentration-time curve (AUC0-24h) of cyclophosphamide. | prexasertib and cyclophosphamide treatment course 1, days 1 and 2
  Cyclophosphamide area under the curve (AUC0-24h) is estimated based on course 1, days 1 and 2 PK samples.
To characterize the systemic clearance (CL) of cyclophosphamide. | prexasertib and cyclophosphamide treatment course 1, days 1 and 2
  Cyclophosphamide systemic clearance (CL) is estimated based on course 1, days 1 and 2 PK samples.
To characterize the area under the concentration-time curve (AUC0-24h) of 4-hydroxy-cyclophosphamide. | prexasertib and cyclophosphamide treatment course 1, days 1 and 2
  4-hydroxy-cyclophosphamide are under the curve AUC0-24h is estimated based on course 1, days 1 and 2 PK samples.
To characterize the area under the concentration-time curve (AUC0-24h) of carboxyethylphosphoramide mustard. | prexasertib and cyclophosphamide treatment course 1, days 1 and 2
  Carboxyethylphosphoramide mustard area under the curve (AUC0-24h) is estimated based on course 1, days 1 and 2. PK samples.
To characterize the area under the concentration-time curve (AUC0-4h) of gemcitabine. | prexasertib and gemcitabine treatment course 1, day 1.
  Gemcitabine area under the curve (AUC0-4h) is estimated based on course 1, day 1 PK samples.
To characterize the systemic clearance (CL) of gemcitabine. | prexasertib and cyclophosphamide treatment course 1, day 1
  Gemcitabine systemic clearance (CL) is estimated based on course 1, day 1 PK samples.
To characterize the area under the concentration-time curve (AUC0-4h) of gemcitabine triphosphate (only at St. Jude Children's Research Hospital). | prexasertib and cyclophosphamide treatment course 1, day 1
  Gemcitabine triphosphate are under the curve AUC0-4h is estimated based on course 1, day 1 PK samples.

CONTACTS AND LOCATIONS:
Overall Officials: Giles W. Robinson, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant de-identified datasets containing the variables analyzed in the published article will be made available (related to the study primary or secondary objectives contained in the publication). Supporting documents such as the protocol, statistical analyses plan, and informed consent are available through the CTG website for the specific study. Data used to generate the published article will be made available at the time of article publication. Investigators who seek access to individual level de-identified data will contact the computing team in the Department of Biostatistics (ClinTrialDataRequest@stjude.org) who will respond to the data request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available at the time of article publication.
Access Criteria: Data will be provided to researchers following a formal request with the following information: full name of requestor, affiliation, data set requested, and timing of when data is needed. As an informational point, the lead statistician and study principal investigator will be informed that primary results datasets have been requested.

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols
- See also: St. Jude Brain Tumor Studies — http://www.stjude.org/research/clinical-trials.html#c671955e2f6ffa4a5f9cd8cf39931465e1f28ef99042a579a1474aa7f29de3b5=2

DOCUMENTS (1):
  • Informed Consent Form (2019-07-10): https://cdn.clinicaltrials.gov/large-docs/69/NCT04023669/ICF_000.pdf